CLINICAL TRIAL: NCT04158583
Title: An Open-Label, Multicenter Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7296682, A CD25-Targeting, T-Regulatory Cell Depleting Antibody in Participants With Advanced and/or Metastatic Solid Tumor
Brief Title: A Study to Evaluate the Safety and Tolerability of RO7296682 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Halted in order to focus on the ongoing combination of RO7296682 with Atezolizumab, evaluated in study BP42595, as a higher likelihood for efficacy is expected in combination with Atezolizumab as compared to the monotherapy setting.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP41188; 2019-002830-35 (EudraCT Number); RG6292 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2019-11-05; First posted 2019-11-12 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumors
Keywords: RG6292

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A: Cohort 1 RO7296682 0.3 mg Q3W (Experimental): Participants with non-small cell lung cancer (NSCLC), melanoma (MEL), head and neck squamous cell carcinoma (HNSCC), ovarian cancer (OvC), triple-negative breast cancer (TNBC), and esophageal carcinoma (EsC) received RO7296682 0.3 milligram (mg) intravenous (IV) infusion on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, every 3 weeks (Q3W). Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 2 RO7296682 1 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 1 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 3 RO7296682 2 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 2 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 4 RO7296682 6 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 6 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 5 RO7296682 18 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 18 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 6 RO7296682 35 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 35 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 7 RO7296682 70 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 70 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 8 RO7296682 100 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 100 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 9 RO7296682 165 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 165 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682
- Part A: Cohort 10 RO7296682 20 mg Q3W (Experimental): Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 20 mg, IV infusion, on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
  Interventions: Drug: RO7296682

INTERVENTIONS:
Drug: RO7296682 — RO7296682 will be administered by the schedules specified in the respective arms.

SUMMARY:
This study was planned to evaluate the safety and tolerability of RO7296682 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
A Phase 1, open-label, dose-escalation study designed to evaluate the safety and tolerability of RO7296682 in participants with advanced and/or metastatic solid tumors. RO7296682 was administered by IV infusion Q3W. This entry-into-human study is divided into a dose-escalation stage (Part A) and a dose expansion stage (Part B).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced and/or metastatic solid tumors who have progressed on all standard therapies, are intolerant to Standard-Of-Care (SOC), and/or are non-amenable to SOC. Participants whose tumors have known sensitizing mutation must have experienced disease progression (during or after treatment) or intolerance to treatment with a respective targeted therapy.
2. Measurable disease according to response evaluation criteria in solid tumors (RECIST) v1.1.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Able to provide the most recent archival tumor tissue samples.
5. Adequate cardiovascular, haematological, liver and renal function.
6. Participants on therapeutic anticoagulation must be on a stable anticoagulant regimen.
7. Women of Childbearing Potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods.
8. Men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods and refrain from donating sperm.

Exclusion Criteria:

1. Pregnancy, lactation, or breastfeeding.
2. Known hypersensitivity to any of the components of RO7296682, including but not limited to hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
3. History or clinical evidence of central nervous system (CNS) primary tumors or metastases.
4. Participants with another invasive malignancy in the last two years.
5. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results.
6. Participants with known active or uncontrolled infection.
7. Positive human immunodeficiency virus (HIV) test at screening.
8. Positive for Hepatitis B and C.
9. Vaccination with live vaccines within 28 days prior to C1D1.
10. Major surgical procedure or significant traumatic injury within 28 days prior to first RO7296682 infusion.
11. Participants with wound healing complications.
12. Dementia or altered mental status that would prohibit informed consent.
13. History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or DRESS (drug rash with eosinophilia and systemic symptoms).
14. Active or history of autoimmune disease or immune deficiency.
15. Prior treatment with checkpoint inhibitors (CPIs) (e.g. anti-CTLA4, anti-PD1, anti-PDL1), immunomodulatory monoclonal antibodies (mAbs) and/or mAb-derived therapies (approved or investigational) is approved.
16. Prior treatment with a CC chemokine receptor 4 (CCR4)-targeting (e.g. mogamulizumab) or a CD25-targeting agent (e.g. basiliximab) is prohibited.
17. Treatment with standard radiotherapy, any chemotherapeutic agent, targeted therapy or treatment with any other investigational drug (defined as treatment for which there is currently no regulatory authority-approved indication) within 28 days or 5 half-lives of the drug (whichever is shorter), prior to the first RO7296882 administration on C1D1.
18. Radiotherapy within the last 4 weeks before start of study drug treatment, with the exception of limited palliative radiotherapy (for which no wash out period is required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria, Australia
- Cliniques Universitaires St-Luc, Brussels, Belgium
- Canada (3):
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Spain (5):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in Part A of the study at 11 centers in Australia, Belgium, Canada, Denmark and Spain from 09 December 2019 to 21 July 2022. The study was terminated before Part B was initiated.
Pre-assignment Details: A total of 76 participants with non-small cell lung cancer (NSCLC), melanoma (MEL), head and neck squamous cell carcinoma (HNSCC), ovarian cancer (OvC), triple-negative breast cancer (TNBC), and esophageal carcinoma (EsC) were enrolled in Part A. No Participants were enrolled in Part B.
Groups:
- Part A: Cohort 1 RO7296682 0.3 mg Q3W: Participants with NSCLC, MEL, HNSCC, OvC, TNBC, and EsC received RO7296682 0.3 mg IV infusion on Day 1 of Cycle 1 (1 cycle=21 days), and at subsequent cycles, Q3W. Participants experiencing toxicities fulfilling the definition of a DLT (e.g: skin toxicities; Grade >=4, IRR; Grade >=4, immune-mediated adverse events; Grade >=4) were discontinued from study treatment.
Period: Overall Study
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Started | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
Pharmacokinetic Population | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 5 | 5 | 6 | 11 | 7 | 4 | 13 | 4 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 3 | 5 | 0 | 1 | 6 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Due To Patient Status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 3 | 4 | 2 | 2 | 4 | 3 | 5 | 2 | 0 | 1
Not completed — Clinical Progression Disease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Clinical Deterioration | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W | Total
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (3.1) | 57.2 (10.9) | 56.8 (17.0) | 56.4 (9.4) | 60.6 (10.0) | 55.4 (9.2) | 60.3 (11.0) | 58.8 (10.3) | 57.0 (14.8) | 59.5 (14.4) | 58.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 7 | 5 | 3 | 8 | 4 | 4 | 4 | 43
  Male | 2 | 2 | 4 | 7 | 3 | 2 | 7 | 2 | 2 | 2 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 6
  Race: White | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 5 | 5 | 5 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 5 | 4 | 6 | 12 | 7 | 5 | 14 | 6 | 6 | 5 | 70
  Ethnicity: Not Stated | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  Ethnicity: Unknown | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) Determined According to The National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From signing of informed consent form (ICF) until last follow-up visit (Up to approximately 2 years 7 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
Participants | 5 | 5 | 6 | 14 | 8 | 5 | 14 | 6 | 6 | 6

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as occurrence of a clinically significant adverse event (AE) from first administration of RO7296682 up to 7 days after second administration of RO7296682. DLTs were defined as following: 1) Hematologic toxicities - Grade 4 neutropenia lasting >=7 days, Grade >=3 febrile neutropenia, Grade 4 thrombocytopenia lasting >=48 hours, Grade 3 thrombocytopenia associated with bleeding episode and Grade 4 anemia 2) Nonhematologic toxicities - Grade 3 nausea, vomiting or diarrhea, Grade >=3 fatigue, Grade 3 arthralgia, fever >40 degree Celsius occurs within 48 hours, Grade >+ laboratory abnormalities, Grade 3 autoimmune thyroiditis or other endocrine abnormalities, Grade 3 tumor flare, Grade 3 transient increase of bilirubin in participants with liver lesions, transaminases (aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) and/or gamma-glutamyl transferase (GGT) and any other RO7296682-related toxicity significant enough to be qualified as DLT.
Time Frame: Up to 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 1

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigators' assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. CR is the disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to < 10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the Baseline sum diameters in the absence of CR.
Time Frame: From treatment initiation until last follow-up visit (Up to approximately 2 years 7 months )
Population: Intent-to Treat (ITT) population included all participants who received at least one dose of RO7296682, and who had at least one baseline and one on-study tumor assessment. Participants who received at least one dose of study drug and discontinued the study because of progression before the first on-study tumor assessment were considered as response-evaluable were included in the efficacy analyses. Participants with missing or no response assessments were classified as not evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
percentage of participants | 0 [0.0 to 52.18] | 0 [0.0 to 52.18] | 0 [0.0 to 45.93] | 0 [0.0 to 23.16] | 0 [0.0 to 36.94] | 0 [0.0 to 52.18] | 0 [0.0 to 21.80] | 0 [0.0 to 45.93] | 0 [0.0 to 45.93] | 0 [0.0 to 45.93]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR defined as the percentage of participants with an overall response of either CR, PR, or stable disease (SD), based on Investigators' assessment using RECIST Version 1.1. CR is defined as disappearance of all target lesions. any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PD is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for (PD). PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline (nadir).
Time Frame: From treatment initiation until last follow-up visit (Up to approximately 2 years 7 months)
Population: ITT population included all participants who received at least one dose of RO7296682, and who had at least one baseline and one on-study tumor assessment. Participants who received at least one dose of study drug and discontinued the study because of progression before the first on-study tumor assessment were considered as response-evaluable were included in the efficacy analyses. Participants with missing or no response assessments were classified as not evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
percentage of participants | 40.0 [5.27 to 85.34] | 20.0 [0.51 to 71.64] | 33.3 [4.33 to 77.72] | 14.3 [1.78 to 42.81] | 37.5 [8.52 to 75.51] | 20.0 [0.51 to 71.64] | 33.3 [11.82 to 61.62] | 33.3 [4.33 to 77.72] | 66.7 [22.28 to 95.67] | 0 [0.0 to 45.93]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first occurrence of a documented objective response to disease progression as determined by the investigator according to RECIST v1.1. or death from any cause, whichever occurs first. Objective response is defined as the percentage of participants having a CR or PR as determined by investigators' assessment of radiographic disease per RECIST v1.1. CR is the disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the SOD of target lesions, taking as reference the Baseline sum diameters in the absence of CR.
Time Frame: From treatment initiation until last follow-up visit (Up to approximately 2 years 7 months)
Population: Participants who received at least one dose of study drug and discontinued the study because of progression before the first on-study tumor assessment were considered as response-evaluable were included in the efficacy analyses. No participants had an objective response, Hence DOR could not be measured.
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: On-Treatment Progression Free Survival (PFS)
Description: The PFS on treatment was defined as the time from study treatment initiation (Cycle 1 Day 1, (1 cycle=21 days) ) to the first occurrence of documented disease progression based on RECIST Version 1.1 Investigator's assessment, or death from any cause, whichever occurred first. For participants who did not have documented progressive disease or death (within 30 days from last study treatment) during the study, PFS was censored at the day of the last tumor assessment. Participants without any post baseline assessments or with all post-baseline assessments having unknown result/response but known to be alive at the clinical cut off for the analysis would be censored at the date of study treatment initiation plus one day.
Time Frame: From treatment initiation until last follow-up visit (Up to approximately 2 years 7 months)
Population: ITT population included all participants who received at least one dose of RO7296682, and who had at least one baseline and one on-study tumor assessment. Participants who received at least one dose of study drug and discontinued the study because of progression before the first on-study tumor assessment were considered as response-evaluable were included in the efficacy analyses.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
days | 59.0 [32.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 59.0 [44.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 43.5 [32.0 to 60.0] | 55.5 [50.0 to 57.0] | 56.5 [15.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 55.0 [26.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 57.0 [51.0 to 63.0] | 58.0 [52.0 to 170.0] | 113.0 [56.0 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 54.0 [39.0 to 57.0]

7. Secondary Outcome: Area Under the Serum Concentration Time Curve (AUC) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: Pharmacokinetic population included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample. Number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms per milliliter(h*μg/mL)
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
hour*micrograms per milliliter(h*μg/mL)
  Cycle 1: number analyzed (Participants) | 4 | 4 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
  Cycle 1 | 12.6 (46.0) | 46.9 (8.7) | 104 (33.4) | 280 (29.5) | 980 (41.1) | 1750 (23.2) | 3940 (29.6) | 5920 (38.8) | 10600 (34.4) | 1040 (22.7)
  Cycle 3/4: number analyzed (Participants) | 2 | 2 | 2 | 13 | 2 | 4 | 6 | 4 | 4 | 3
  Cycle 3/4 | 26.5 (52.4) | 39.8 (63.5) | 109 (7.2) | 359 (53.6) | 1140 (26.3) | 2510 (19.0) | 5110 (55.1) | 8070 (49.6) | 11900 (37.7) | 1460 (45.2)

8. Secondary Outcome: Minimum Serum Concentration (Cmin) of RO7296682
Time Frame: Cycles 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 3 | 2 | 2 | 13 | 2 | 4 | 7 | 4 | 5 | 4
μg/mL | NA (NA) — Geometric mean and geometric coefficient of variation could not be calculated due to insufficient number of participants with events. | 0.0546 (NA) — Geometric coefficient of variation could not be calculated due to insufficient number of participants with events. | 0.0858 (8.4) | 0.265 (0.0519) | 1.02 (32.6) | 1.40 (29.5) | 4.77 (72.0) | 5.83 (126.6) | 11.4 (47.3) | 1.11 (51.8)

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
μg/mL
  Cycle 1 | 0.0718 (26.9) | 0.256 (16.1) | 0.505 (34.3) | 1.79 (57.5) | 5.38 (31.3) | 9.80 (29.1) | 22.4 (25.9) | 38.2 (26.7) | 75.9 (46.2) | 7.46 (30.6)
  Cycle 3/4: number analyzed (Participants) | 3 | 2 | 2 | 13 | 2 | 4 | 7 | 4 | 5 | 4
  Cycle 3/4 | 0.107 (51.7) | 0.277 (8.4) | 0.727 (42.4) | 2.58 (80.2) | 5.22 (16.3) | 14.0 (24.2) | 24.0 (32.9) | 41.8 (18.6) | 72.8 (33.7) | 7.24 (58.3)

10. Secondary Outcome: Total Clearance (CL) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
milliliter per hour (mL/h)
  Cycle 1: number analyzed (Participants) | 4 | 4 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
  Cycle 1 | 23.9 (46.0) | 21.3 (8.7) | 19.3 (33.4) | 21.4 (29.5) | 18.4 (41.1) | 20.0 (23.2) | 17.8 (29.6) | 16.9 (38.8) | 15.5 (34.4) | 19.2 (22.7)
  Cycle 3/4: number analyzed (Participants) | 2 | 2 | 2 | 13 | 2 | 4 | 6 | 4 | 4 | 3
  Cycle 3/4 | 20.7 (37.1) | 25.2 (63.5) | 18.3 (7.2) | 16.7 (53.6) | 15.8 (26.3) | 13.9 (19.0) | 10.9 (65.1) | 12.4 (49.6) | 13.9 (37.7) | 13.7 (45.2)

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
milliliter (mL)
  Cycle 1: number analyzed (Participants) | 4 | 4 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
  Cycle 1 | 7480 (61.4) | 5840 (20.1) | 7570 (60.8) | 6150 (23.8) | 5500 (34.9) | 6920 (38.3) | 6140 (29.2) | 5020 (29.0) | 4510 (23.5) | 5650 (16.8)
  Cycle 3/4: number analyzed (Participants) | 2 | 2 | 2 | 12 | 2 | 4 | 6 | 4 | 4 | 3
  Cycle 3/4 | 7340 (24.6) | 5410 (14.5) | 5200 (37.6) | 4710 (34.1) | 5520 (25.5) | 4550 (40.6) | 5030 (18.0) | 3850 (20.6) | 4060 (48.6) | 5240 (18.5)

12. Secondary Outcome: Terminal Half-Life (T1/2) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
hours
  Cycle 1: number analyzed (Participants) | 4 | 4 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
  Cycle 1 | 286 [68.3 to 352] | 213 [135 to 243] | 382 [168 to 410] | 204 [130 to 292] | 241 [94.8 to 367] | 264 [209 to 336] | 232 [128 to 463] | 199 [129 to 359] | 198 [176 to 219] | 242 [128 to 270]
  Cycle 3/4: number analyzed (Participants) | 3 | 2 | 2 | 12 | 2 | 4 | 6 | 4 | 4 | 3
  Cycle 3/4 | 244 [241 to 246] | 170 [89.3 to 252] | 206 [157 to 255] | 215 [93.1 to 318] | 265 [169 to 361] | 231 [171 to 356] | 356 [152 to 642] | 265 [118 to 309] | 267 [105 to 281] | 226 [219 to 489]

13. Secondary Outcome: Time of Maximum Concentration (Tmax) of RO7296682
Time Frame: Cycles 1, and 3 or 4 (Cycle length = 21 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 13 | 6 | 5 | 15 | 6 | 6 | 6
hours
  Cycle 1 | 6.5 [3.92 to 7.73] | 4.05 [0 to 4.33] | 5.31 [3.67 to 7.00] | 4.08 [3.97 to 46.43] | 5.36 [4.07 to 6.83] | 4.08 [4.00 to 7.23] | 4.20 [2.00 to 6.72] | 4.20 [4.02 to 6.83] | 4.07 [2.00 to 6.73] | 6.68 [2.00 to 21.25]
  Cycle 3/4: number analyzed (Participants) | 3 | 2 | 2 | 13 | 2 | 4 | 7 | 4 | 5 | 4
  Cycle 3/4 | 1.00 [0.98 to 3.63] | 2.31 [1.12 to 3.50] | 3.52 [3.50 to 3.53] | 1.08 [0.58 to 23.67] | 1.14 [1.08 to 1.20] | 3.83 [3.58 to 24.83] | 1.05 [0.68 to 22.42] | 2.38 [1.07 to 4.65] | 1.02 [1.00 to 3.57] | 21.57 [1.07 to 49.32]

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) During the Study Relative to the Prevalence of ADA at Baseline
Time Frame: Predose on Day 1 of each 21-day and subsequent cycles up to end of study (Up to approximately 2 years 7 months)
Population: Immunogenicity analyses population included all participants with at least one ADA assessment, irrespective of whether or not the participant received any treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Treatment-induced Changes in Treg Levels in Blood and/or Tumor as Compared to Baseline
Time Frame: Baseline and at Cycle 1 Day 4 (Cycle length = 21 days)
Population: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not. Number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percent cells per microliter (cells/µL)
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
percent cells per microliter (cells/µL)
  %CD4 Treg: Baseline: number analyzed (Participants) | 4 | 4 | 5 | 11 | 7 | 4 | 12 | 5 | 6 | 5
  %CD4 Treg: Baseline | 1.61 (0.36) | 2.77 (1.31) | 1.94 (1.54) | 2.39 (2.20) | 1.65 (1.17) | 3.40 (0.25) | 2.65 (1.48) | 1.84 (0.64) | 1.92 (1.51) | 2.20 (1.78)
  %CD4 Treg: Change from Baseline at Cycle 1 Day 4: number analyzed (Participants) | 4 | 4 | 5 | 10 | 6 | 3 | 11 | 5 | 5 | 4
  %CD4 Treg: Change from Baseline at Cycle 1 Day 4 | 0.18 (2.15) | -1.22 (0.88) | -1.17 (1.33) | -1.71 (1.95) | -0.79 (2.29) | -3.02 (0.56) | -2.62 (1.38) | -1.33 (0.61) | -1.98 (1.04) | -1.28 (1.10)

16. Secondary Outcome: Treatment-induced Changes in Treg/Teff (T-regulatory Cell; T-effector Cell) Ratio in Blood and/or Tumor as Compared to Baseline
Time Frame: Baseline and at Cycle 1 Day 4 (Cycle length = 21 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
Number analyzed (Participants) | 5 | 5 | 6 | 14 | 8 | 5 | 15 | 6 | 6 | 6
ratio
  Treg/Teff Ratio: Baseline: number analyzed (Participants) | 4 | 4 | 5 | 11 | 7 | 4 | 12 | 5 | 6 | 5
  Treg/Teff Ratio: Baseline | 0.05 (0.04) | 0.06 (0.04) | 0.10 (0.09) | 0.06 (0.05) | 0.05 (0.04) | 0.10 (0.06) | 0.11 (0.10) | 0.07 (0.07) | 0.04 (0.04) | 0.05 (0.05)
  Treg/Teff Ratio: Change from Baseline at Cycle 1 Day 4: number analyzed (Participants) | 4 | 4 | 5 | 10 | 6 | 3 | 11 | 6 | 5 | 3
  Treg/Teff Ratio: Change from Baseline at Cycle 1 Day 4 | 12.50 (51.90) | 19.0 (131.90) | 30.0 (53.35) | 52.30 (113.88) | -9.17 (98.55) | -5.33 (33.86) | -14.64 (67.96) | -12.33 (104.22) | 26.00 (79.05) | -121.00 (108.75)

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years 7 months
Description: Safety population included all participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | Part A: Cohort 1 RO7296682 0.3 mg Q3W | Part A: Cohort 2 RO7296682 1 mg Q3W | Part A: Cohort 3 RO7296682 2 mg Q3W | Part A: Cohort 4 RO7296682 6 mg Q3W | Part A: Cohort 5 RO7296682 18 mg Q3W | Part A: Cohort 6 RO7296682 35 mg Q3W | Part A: Cohort 7 RO7296682 70 mg Q3W | Part A: Cohort 8 RO7296682 100 mg Q3W | Part A: Cohort 9 RO7296682 165 mg Q3W | Part A: Cohort 10 RO7296682 20 mg Q3W
All-Cause Mortality (participants affected / at risk) | 3/5 | 4/5 | 5/6 | 7/14 | 5/8 | 4/5 | 10/15 | 4/6 | 1/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/5 | 0/6 | 7/14 | 3/8 | 0/5 | 5/15 | 0/6 | 1/6 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 6/6 | 14/14 | 8/8 | 5/5 | 14/15 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1 RO7296682 0.3 mg Q3W (N=5) | Part A: Cohort 2 RO7296682 1 mg Q3W (N=5) | Part A: Cohort 3 RO7296682 2 mg Q3W (N=6) | Part A: Cohort 4 RO7296682 6 mg Q3W (N=14) | Part A: Cohort 5 RO7296682 18 mg Q3W (N=8) | Part A: Cohort 6 RO7296682 35 mg Q3W (N=5) | Part A: Cohort 7 RO7296682 70 mg Q3W (N=15) | Part A: Cohort 8 RO7296682 100 mg Q3W (N=6) | Part A: Cohort 9 RO7296682 165 mg Q3W (N=6) | Part A: Cohort 10 RO7296682 20 mg Q3W (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1 RO7296682 0.3 mg Q3W (N=5) | Part A: Cohort 2 RO7296682 1 mg Q3W (N=5) | Part A: Cohort 3 RO7296682 2 mg Q3W (N=6) | Part A: Cohort 4 RO7296682 6 mg Q3W (N=14) | Part A: Cohort 5 RO7296682 18 mg Q3W (N=8) | Part A: Cohort 6 RO7296682 35 mg Q3W (N=5) | Part A: Cohort 7 RO7296682 70 mg Q3W (N=15) | Part A: Cohort 8 RO7296682 100 mg Q3W (N=6) | Part A: Cohort 9 RO7296682 165 mg Q3W (N=6) | Part A: Cohort 10 RO7296682 20 mg Q3W (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid skin dryness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 5 (7) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (3) | 4 (5) | 0 (0) | 5 (10) | 1 (1) | 2 (2) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 1 (2) | 0 (0) | 2 (2) | 2 (3) | 2 (3) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 5 (11) | 0 (0) | 2 (2) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 6 (9) | 0 (0) | 3 (3) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 1 (1) | 3 (4) | 7 (7) | 3 (4) | 1 (1) | 4 (4)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (4) | 5 (9) | 3 (5) | 2 (2) | 4 (9) | 1 (2) | 0 (0) | 4 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04158583/Prot_SAP_000.pdf